CLINICAL TRIAL: NCT05599919
Title: A Randomized, Double-blind, Parallel Arm, Multicenter Study To Evaluate The Efficacy And Safety Of Nitric Oxide Nasal Spray Combined With Standard Supportive Care In Adult Non-hospitalized Patients With COVID-19.
Brief Title: Nitric Oxide Nasal Spray (NONS) To Treat and Prevent the Exacerbation of Infection in Individuals With Mild COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanotize Research and Development corp. (Industry)
Collaborators: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GPL/CT/2021/004/III
Record Dates: First submitted 2022-05-03; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-02

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Nitric Oxide; Nasal Sprays

STUDY DESIGN:
Intervention Model Description: The primary objective of this study is to evaluate the efficacy of Nitric Oxide Nasal Spray combined with standard supportive care compared with standard supportive care alone in adult subjects with COVID-19 not requiring hospitalization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with COVID-19 (confirmed by RT-PCR), not requiring hospitalization (Active Comparator): Nitric oxide releasing solution delivered up to 3 times daily
  Interventions: Drug: Nitric Oxide
- COVID-19 symptoms (Placebo Comparator): saline delivered up to 3 times daily morning, mid-day, and evening. Maximum volume delivered: 0.56 mL Saline @ 0.9%
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — The Sponsor designed a dual chamber nasal spray bottle for NORS administration. Components are mixed from two chambers to create the final NO-producing formulation. The liquid contains NO at 0.11 ppm*hour, which acts as a viricidal agent. Instructions for storing, preparing, and administering the study treatment will be provided to participants.
  Other Names: Nasal Spray

SUMMARY:
Primary:

The primary objective of this study is to evaluate the efficacy of Nitric Oxide Nasal Spray combined with standard supportive care compared with standard supportive care alone in adult subjects with COVID-19 not requiring hospitalization

Secondary:

The secondary objective is to evaluate the safety and tolerability of Nitric Oxide Nasal Spray combined with standard supportive care compared with standard supportive care alone in adult subjects with COVID-19 not requiring hospitalization.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multi-center, parallel arm, clinical study evaluating the efficacy and safety of Nitric Oxide Nasal Spray with standard supportive care vs standard supportive care alone in patients with COVID-19 not requiring hospitalization.

306 eligible patients will be randomized in a 1:1 ratio into 2 groups: one group will receive Nitric Oxide Nasal Spray (NONS) along with standard supportive care and the control group will receive standard supportive care along with placebo of NONS. Standard supportive care will be provided in accordance with latest guidelines issued by Ministry of Health and family welfare; Government of India. Treatment duration is 7 days (up to Day 8 visit) and the total study duration will be maximum for 18 days from randomization (up to Day 19 visit). Viral load will be estimated on Day 1 (baseline), Day 2 (post-24 hours of dosing), Day 3 (post 48 hours of dosing), Day 4 (post 72 hours of dosing) and Day 8. Patients may be detained in a facility to facilitate protocol assessments for first 7 days or may be treated at home based on investigator discretion. Subjects who are treated at home will visit the study center on Day 1, 4, and 8 for study assessments and Day 2 visit (and swab sample collection for visit 2) will be conducted at home. Day 3 will be laboratory visit only for collection of swab from both sides in the nose for RT-PCR. If subjects are not able to visit the study center on any of the days, telephonic or video-conference and home based assessments can be conducted.

On Day 1 (screening and randomization), written informed consent will be obtained from subjects with symptoms of COVID-19 and having symptom onset within 48 hours before consent. After informed consent, following activities will be conducted: detailed clinical history and physical examination, vaccination status, vital signs, SpO2 measurement, 12-lead ECG, chest x-ray, eligibility assessment and blood and urine collection for laboratory assessments (including C-Reactive Protein). Rapid positive result for COVID-19 antigen will be randomized. Subjects with negative result for COVID-19 antigen will be considered as screen failure. Only swab from both sides in the nose will be taken as per the standard procedure for quantitative and qualitative RT-PCR assessments. If the result of qualitative RT-PCR of swab sample collected during screening is negative, subject will be withdrawn from the study. After screening procedures subjects will be randomized to one of the two treatment arms and investigational product (IP) will be dispensed. After training on nasal spray administration, first dose will be self-administered under supervision. Standard supportive care will be provided to all the subjects during the study.

On Day 2, 3 and 4 swab from both sides in the nose will be taken for quantitative and qualitative RT-PCR. On Day 2 and 4 following study procedures will be conducted: adverse event review, concomitant medication review, IP compliance review, SpO2, vital signs. On Day 4 a chest x-ray or CT scan will be done (choice between x-ray and CT scan at Day 4 will be based on investigator discretion). Only for subjects who are not able to visit the site can conduct chest x-ray or CT scan at nearby facility. Day 3 will be a Laboratory visit during which swab will be collected from nose for RT-PCR. On Day 8 subject will visit the study site and following activities will be performed: adverse event review, concomitant medication review, IP compliance review, SpO2, vital signs, physical examination, 12-lead ECG, blood and urine collection for laboratory assessments. Swab from both sides in the nose will be taken for qualitative and quantitative RT-PCR assessment, and IP will be retrieved. Qualitative and quantitative RT-PCR assessments will be done in all subjects on days 2, 3 and 4, irrespective of RT-PCR result (positive or negative) on days 2 and 3. Subjects who have negative result of qualitative RT-PCR (RT-PCR negative) at Day 4, RT-PCR (both qualitative and quantitative) will not be done on Day 8 and rest of the assessments as per visit schedule for Day 8 will be conducted. Visit 5 will be conducted on Day 19 ± 2 days or any time between Day 8 and Day 19, if the subject's COVID-19 symptom status and RT-PCR result becomes negative. Visit 5 will be a telephonic visit or clinic visit. During visit 5, history of adverse events and concomitant medication will be taken and in case of adverse event a clinic visit can be performed based on investigator's discretion for detailed assessments or additional tests. For subjects who are RT-PCR positive on Day 8, standard of care will be continued and swab from both sides in the nose will be collected at visit 5 for qualitative RT-PCR assessment. On Day 1, 2, 4, and 8; and at visit 5 information about immediate contacts and their COVID-19 status will be collected. During the study, following events will be recorded: first time use of high flow supplemental oxygen, hospitalization for treatment purposes (COVID-19 related), non-invasive ventilation, mechanical ventilation, and extracorporeal membrane oxygenation and symptom scales. Methemoglobin will be measured non-invasively in a subset of patients on Day 1 [before randomization (baseline), and 5 minutes after administration of first dose of NONS], Day 2, Day 4 and Day 8. Subject diary will be used to record information related to adverse events, use of concomitant medications and study drug compliance. Subject diary will be dispensed at screening/randomization visit (visit 1) and retrieved at Day 8 (visit 4). Subjects will record their health status and COVID-19 related symptoms daily during the study participation using the subject diary. Investigator will record the score on the WHO Progression Scale at visits 1, 2, 3, 4 and 5. After Day 8 visit, additional qualitative RT-PCR tests can be conducted as unscheduled investigations in subjects who are RT-PCR positive on Day 8. Subjects whose baseline COVID-19 symptoms have resolved by Day 8 and whose RT-PCR is negative by Day 8, will not undergo any further assessment (including visit 5) and their study participation will be considered as complete. For subjects whose baseline COVID-19 symptoms are present at Day 8 and/or whose RT-PCR is positive at Day 8 will be continued in the study till maximum of Day 19. Between Day 8 and Day 19 on or after the day the subject becomes RT-PCR negative and has baseline COVID-19 symptoms resolved, visit 5 can be conducted and subject's study participation can be considered complete. All subjects study participation, irrespective of RT-PCR and symptom status will end on maximum of Day 19±2 days (visit 5).

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be entered into the randomized treatment in the study:

1. Voluntarily participating in the clinical study; fully understanding and being fully informed of the study and having signed the Informed Consent Form (ICF); willingness and capability to complete all the study procedures
2. Age 18-65 years (inclusive) at the time of signing ICF
3. Patients with laboratory confirmation of infection with SARS-CoV-2 by positive Rapid Antigen Test for SARS-CoV-2 at screening.
4. Recent onset (within 48 hours of time of consent) symptoms of mild COVID-19 with oxygen saturation (SpO2 > 94 %) and respiratory rate < 24 breaths/min. Any of the COVID-19 like symptoms including fever, cough, sore throat, malaise, headache, nasal congestion, muscle pain, gastrointestinal symptoms, lack of taste or smell without shortness of breath or dyspnea; (the maximum permitted difference in the time of onset of symptoms and the time of consent is 48 hours)
5. For female subjects: evidence of post-menopause, or, for pre-menopause subjects, negative pretreatment urine pregnancy test
6. Eligible subjects of child-bearing age (female or male with female partner of childbearing age) must agree to take effective contraceptive measures (including hormonal contraception, barriermethods or abstinence) with his/her partner during the study period and for at least 7 days following the last study treatment.
7. Not participating in any other interventional drug clinical studies before completion of the present study.

Exclusion Criteria:

A subject who meets any of the following criteria must not be entered into the randomized treatment in the study:

1. Where, in the opinion of the investigator, participation in this study will not be in the best interest of the subject, or any other circumstances that prevent the subject from participating in the study safely
2. Subjects with infection requiring oxygen support, invasive or non-invasive ventilator support, extracorporeal membrane oxygenation (ECMO) or shock requiring vasopressor support.
3. Current known pneumonia based on x-ray or computed tomography (CT) scan or history of pneumonia within 3 months before screening.
4. Requiring hospitalization for the treatment of COVID-19
5. Subjects who have received any dose of vaccine for COVID-19
6. Prolonged QT, defined as QTcF ≥ 450 milliseconds for men and as QTcF ≥ 470 milliseconds for women
7. History of known severely reduced left ventricular (LV) function (Ejection fraction < 30 %)
8. Requires ICU care for management of ongoing clinical status.
9. Known allergy or hypersensitivity to Nitric Oxide Nasal Spray.
10. History of known severe renal impairment [creatinine clearance (CrCl) < 30 mL/min] or having received continuous renal replacement therapy, hemodialysis or peritoneal dialysis;
11. Asthma, allergic rhinitis or chronic obstructive lung disease
12. Psychiatric disease that is not well controlled (controlled defined as stable on a regimen for more than one year).
13. Pregnant or lactating women;
14. Having used Nitric Oxide Nasal Spray or participated in any other interventional drug clinical study within 30 days prior to first dose of study drug.
15. Subjects who have received hydroxychloroquine within 7 days before screening or subjects who require hydrochloroquine treatment.
16. Subjects who have received intranasal medication/treatment within 7 days before screening or subjects who require use of any intranasal medication.
17. Subjects who have received medications with antiviral effect such as remdesivir, favipiravir, oseltamivir, ivermectin or inhaled corticosteroids within 7 days before screening or subjects who require use of any of these medications
18. Subjects using nitric oxide donor agents such as prilocaine, sodium nitroprusside and nitroglycerine Duration of study participation: The anticipated maximum total study duration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the efficacy of Nitric Oxide Nasal Spray combined with standard supportive care compared with standard supportive care alone in adult subjects with COVID-19 not requiring hospitalization | 8 days
  Change from baseline in log viral load

SECONDARY OUTCOMES:
The secondary objective is to evaluate the safety and tolerability of Nitric Oxide Nasal Spray combined with standard supportive care compared with standard supportive care alone in adult subjects with COVID-19 not requiring hospitalization. | 18 days
  Number of adverse events, pain, discomfort or discontinuations of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Keith Moore, PHARMD, Study Director — kmoore@sanotize.com
Locations (21):
- India (21):
  - Ishwar Institute & Hospital, Aurangabad
  - MGM Medical College & Hospital, Aurangabad
  - Bangalore Medical College and Research Institute, Bangalore
  - Hindusthan Hospital, Coimbatore
  - Marwari Hospital, Guwahati
  - St.Theresas Hospital, Hyderabad
  - Aster Prime Hospital, Hyderabad
  - Renova Neelima Hospitals, Hyderabad
  - Prakash Institute of Medical Sciences & Research, Islāmpur
  - Maharaja Agrasen Superspeciality Hospital, Jaipur
  - Pharmacology Dept. CPR Hospital Campus, Town Hall,, Kolhāpur
  - C K Birla Hospitals, The Calcutta Medical Research Institute, Kolkata
  - Peerless Hospitex Hospital And Research Centre Limited, Kolkata
  - CSI Medical College and Hospital, Kolkata
  - Malabar Medical College Hospital and Research Centre, Kozhikode
  - Orchid Specialty Hospital, Lohgaon
  - St. Georges Hospital, Mumbai
  - Dr Rahul Kodgule, Mumbai
  - Government Medical College and Hospital Nagpur, Nagpur
  - All India Institute of Medical Sciences, Nagpur
  - Lifepoint Multispeciality Hospital, Pune